CLINICAL TRIAL: NCT00916435
Title: Prospective Observational Study of the ICD Intracardiac Electrograms for Prediction of Ventricular Tachyarrhythmias and Congestive Heart Failure
Brief Title: Study of the Implantable Cardioverter Defibrillator (ICD) Intracardiac Electrograms
Acronym: ICD-EGMs
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Larisa Tereshchenko, Instructor of Medicine, Johns Hopkins University
Other Study IDs: 1K99HL094665-01 (in review)
Record Dates: First submitted 2009-06-08; First posted 2009-06-09 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Congestive Heart Failure; Sudden Cardiac Death; Arrhythmia; Cardiomyopathies
Keywords: Arrhythmia; Cardiac Arrest; Cardiomyopathy; Heart Failure
MeSH Terms: conditions — Heart Failure; Death, Sudden, Cardiac; Arrhythmias, Cardiac; Cardiomyopathies; Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether waveforms of the intracardiac electrograms, acquired through an ICD, can be used:

* to predict malignant ventricular arrhythmias, requiring appropriate ICD therapies, and
* to predict progression of heart failure in patients with ICD.

ELIGIBILITY:
Inclusion Criteria:

* history of acute MI at least 4 weeks old
* non-ischemic LV dysfunction for at least 9 months
* who have an EF < or = to 35%
* who was resuscitated from sudden cardiac arrest (ventricular tachyarrhythmia)
* undergone implantation of an FDA-approved ICD for primary or secondary prevention of SCD

Exclusion Criteria:

* inability or unwillingness to provide valid informed consent
* pregnancy
* any condition other than cardiac disease that was associated with a high likelihood of death during 1 year after enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic or non-ischemic cardiomyopathy undergoing ICD implantation for primary or secondary prevention of sudden cardiac death
Sampling Method: Probability Sample
Enrollment: 630 (Actual)
Dates: Start 2005-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
sustained ventricular tachycardia with appropriate ICD therapies (either shock or ATP) | from enrollment up to 72 months

SECONDARY OUTCOMES:
Composite heart failure outcome (HF hospitalization, HF death, heart transplant) | from enrollment up to 72 months
All-cause mortality | from enrollment up to 72 months

CONTACTS AND LOCATIONS:
Overall Officials: Larisa G Tereshchenko, MD, PhD, Principal Investigator — Johns Hopkins University; Ronald D Berger, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri

REFERENCES:
- [Result] Tereshchenko LG, Fetics BJ, Domitrovich PP, Lindsay BD, Berger RD. Prediction of ventricular tachyarrhythmias by intracardiac repolarization variability analysis. Circ Arrhythm Electrophysiol. 2009 Jun;2(3):276-84. doi: 10.1161/CIRCEP.108.829440. Epub 2009 Mar 6. PMID 19808478
- [Result] Tereshchenko LG, Fetics BJ, Berger RD. Intracardiac QT variability in patients with structural heart disease on class III antiarrhythmic drugs. J Electrocardiol. 2009 Nov-Dec;42(6):505-10. doi: 10.1016/j.jelectrocard.2009.07.011. Epub 2009 Aug 22. PMID 19700170
- [Result] Tereshchenko LG, Faddis MN, Fetics BJ, Zelik KE, Efimov IR, Berger RD. Transient local injury current in right ventricular electrogram after implantable cardioverter-defibrillator shock predicts heart failure progression. J Am Coll Cardiol. 2009 Aug 25;54(9):822-8. doi: 10.1016/j.jacc.2009.06.004. PMID 19695461
- [Result] Stempniewicz P, Cheng A, Connolly A, Wang XY, Calkins H, Tomaselli GF, Berger RD, Tereshchenko LG. Appropriate and inappropriate electrical therapies delivered by an implantable cardioverter-defibrillator: effect on intracardiac electrogram. J Cardiovasc Electrophysiol. 2011 May;22(5):554-60. doi: 10.1111/j.1540-8167.2010.01958.x. Epub 2010 Nov 18. PMID 21087331
- [Result] Oosterhoff P, Tereshchenko LG, van der Heyden MA, Ghanem RN, Fetics BJ, Berger RD, Vos MA. Short-term variability of repolarization predicts ventricular tachycardia and sudden cardiac death in patients with structural heart disease: a comparison with QT variability index. Heart Rhythm. 2011 Oct;8(10):1584-90. doi: 10.1016/j.hrthm.2011.04.033. Epub 2011 May 10. PMID 21699842
- [Result] Tereshchenko LG, Henrikson CA, Stempniewicz P, Han L, Berger RD. Antiarrhythmic effect of reverse electrical remodeling associated with cardiac resynchronization therapy. Pacing Clin Electrophysiol. 2011 Mar;34(3):357-64. doi: 10.1111/j.1540-8159.2010.02974.x. Epub 2010 Nov 22. PMID 21091740
- [Result] Chen X, Tereshchenko LG, Berger RD, Trayanova NA. Arrhythmia risk stratification based on QT interval instability: an intracardiac electrocardiogram study. Heart Rhythm. 2013 Jun;10(6):875-80. doi: 10.1016/j.hrthm.2013.02.014. Epub 2013 Feb 13. PMID 23416373
- [Result] Das D, Han L, Berger RD, Tereshchenko LG. QT variability paradox after premature ventricular contraction in patients with structural heart disease and ventricular arrhythmias. J Electrocardiol. 2012 Nov-Dec;45(6):652-7. doi: 10.1016/j.jelectrocard.2012.07.016. Epub 2012 Sep 17. PMID 22995383
- [Result] Baumert M, Kabir MM, Dalouk K, Henrikson CA, Tereshchenko LG. VV' Alternans Triplets on Near-Field ICD Intracardiac Electrogram is Associated with Mortality. Pacing Clin Electrophysiol. 2015 May;38(5):547-57. doi: 10.1111/pace.12594. Epub 2015 Mar 9. PMID 25752990
- [Result] Guduru A, Lansdown J, Chernichenko D, Berger RD, Tereshchenko LG. Longitudinal changes in intracardiac repolarization lability in patients with implantable cardioverter-defibrillator. Front Physiol. 2013 Aug 12;4:208. doi: 10.3389/fphys.2013.00208. eCollection 2013. PMID 23964242
- [Result] Tereshchenko LG, McCabe A, Han L, Sur S, Huang T, Marine JE, Cheng A, Spragg DD, Sinha S, Calkins H, Stein K, Tomaselli GF, Berger RD. Intracardiac J-point elevation before the onset of polymorphic ventricular tachycardia and ventricular fibrillation in patients with an implantable cardioverter-defibrillator. Heart Rhythm. 2012 Oct;9(10):1594-602. doi: 10.1016/j.hrthm.2012.06.036. Epub 2012 Jun 29. PMID 22750217